CLINICAL TRIAL: NCT07212062
Title: A Phase II, Randomized, Double-Blind, Placebo Controlled Study to Evaluate the Sfatey and Tolerability of X/T+X-EC vs. Placebo in Participants With Alzheimer's Disease Currently Treated With Lecanemab.
Brief Title: The Purpose of This Study is to Evaluate the Safety and Tolerability of X/T+X-EC in Participants With Alzheimer's Disease Who Are Currently Treated With Lecanemab.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neurology Office of South Florida (Network)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN012-0117; CN012-0117 (Other Grant/Funding Number: Bristol-Myers Squibb); CN012-0117 (Other: Neurology Offices of South Florida (NOSFL))
Record Dates: First submitted 2025-09-22; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Alzheimers Disease
Keywords: Alzheimers Disease; Lecanemab
MeSH Terms: conditions — Alzheimer Disease | interventions — lecanemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A- Lecanemab + X/T + X-EC (Active Comparator): Participants will receive the active drug as well as their current Lecanemab treatment.
  Interventions: Drug: X/T + X-EC; Drug: Lecanemab 10 mg/kg
- Arm B- Lecanemab + Placebo (Placebo Comparator): Participants will receive the non-active drug/placebo as well as their current Lecanemab treatment.
  Interventions: Drug: Placebo; Drug: Lecanemab 10 mg/kg

INTERVENTIONS:
Drug: X/T + X-EC — Xanomeline and Trospium Chloride Capsules
  Arms: Arm A- Lecanemab + X/T + X-EC
Drug: Placebo — Placebo
  Arms: Arm B- Lecanemab + Placebo
Drug: Lecanemab 10 mg/kg — Participants will continue their current Lecanemab infusions while in the study receiving the study drug or placebo.

SUMMARY:
The goal of the trial is to see if the Safety and Tolerability of X/T+X/T-EC combined with currently treated Lecanemab participants with Alzheimer's Disease compared with placebo. This is a 32 week study (4 weeks of screening,24 weeks of treatment and 4 weeks of safety follow up)

DETAILED DESCRIPTION:
Phase II, randomized, double-blind, placebo-controlled study to evaluate the safety and tolerability of X/T+X-EC vs. placebo in participants with Alzheimer's Disease currently treated with Lecanemab. 32 week study. 60 participants (60-85 years of age), 3 US sites. A caregiver/LAR will be utilized for each participant. LAR must be knowledgeable of the participant and spends no less than 10 hours per week with them. Participants must have received treatment with commercially available Lecanemab and must have completed at least 14 infusions prior to screening. Eligible participants will continue with their treatment of Lecanemab. If qualified for the study, the participants will be randomized to either the study drug provided X/T+X-EC or placebo. The radnomization will be performed by the RTSM system.

ELIGIBILITY:
Inclusion Criteria:1. Participants or their legally acceptable representative (LAR, see Appendix 1) must be able and willing to sign and date an IRB/IEC-approved written informed consent form ICF in accordance with regulatory, local, and institutional guidelines. This ICF must be obtained before performing any protocol-related procedures that are not part of normal patient care. Participant must be fluent in the language of the ICF to consent.

Type of Participant and Target Disease Characteristics 2. A diagnosis of AD

1. A confirmed clinical diagnosis of Alzheimer's disease and AD pathology verified by a Health Authority-approved assay. Participants must have received treatment with commercially available Lecanemab (10 mg/kg IV every two weeks) and must have completed at least 14 infusions prior to screening.

   3. BMI within 18 to 35 kg/m2 inclusive. 4. MMSE score 16-24 (inclusive) at screening; 5. Historical MRI prior to 14th infusion of Leqembi®. 6. Participant has a stable living environment for at least 6 weeks prior to screening. Participants are eligible if they are in nursing homes, assisted living facilities, memory care facilities, or living at home.

   7. The participant has sufficient verbal ability to satisfactorily comply with the study procedures (corrective measures such as hearing aids and reading glasses are allowed, if necessary) and is willing and able to attend clinic visits. Participants who use wheelchairs or other ambulatory assistive devices are permitted to enter this study.

   8. Caregiver/study partner must be willing to comply with scheduled visits and protocol standards. In addition; the caregiver/study partner must be in contact with the participant frequently enough to accurately report on the participant's symptoms and on participant's adherence to the study drug schedule, in the investigator's opinion. The caregiver/study partner must be fluent in the local language in which the study assessment will be conducted. The caregiver/study partner must agree to participate in study assessments and provide written consent to participate in the study.

   9. The participant must be willing and able to discontinue all prohibited concomitant medications to meet protocol washout and medication stability requirements before randomization. Investigators should not withdraw a participant's prohibited medication for the purpose of enrolling them into the study unless discontinuation of the medication is deemed to be clinically appropriate (e.g., symptoms are not well-controlled, or the participant cannot tolerate the current medication).

   10. In premorbid state, participant had sufficient literacy and arithmetic proficiency to allow completion of the cognitive assessments.

Age of Participant 11. Participant must be 60 to 85 years, inclusive, at the time of signing the ICF.

12. Female (as assigned at birth) participants who are not of childbearing potential (as defined in Appendix 3) must have documented proof. Documentation can be obtained from the site personnel's review of the participant's medical records, medical examination, or medical history interview.

1. IOCBP must have a negative highly sensitive pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of study intervention.
2. IOCBP must agree to follow instructions for method(s) of contraception as described below and included in the ICF. IOCBP are permitted to use hormonal contraceptive methods (as described in Appendix 3).

Note: 1) If a urine test cannot be confirmed as negative (e.g., an ambiguous result), the participant must be excluded from participation if a repeat serum pregnancy result is positive. 2) The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to potentially decrease the risk for inclusion of an individual with an undetected pregnancy. 3) Individuals who are not of childbearing potential are exempt from contraceptive requirements.

13. A female (as assigned at birth) is eligible to participate if she is not pregnant or breastfeeding and at least 1 of the following conditions applies:

• Is not an IOCBP OR

• Is an IOCBP and using a contraceptive method that is highly effective (with a failure rate of < 1% per year), preferably with user independent methods as described in Appendix 3, during the intervention period and for at least 16 days after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction for the same period.

14. Male participants should maintain their usual practice regarding contraception (if any); however, no specific or additional contraceptive measures are required.

Prior/Concomitant Therapy (See Appendix 4 for complete list of Permitted Concomitant Therapy) 15. If receiving an approved symptomatic AD treatment such as AchEIs or NMDA antagonist (memantine), or both, for AD, participants must be on a stable dose for at least 12 weeks prior to screening and agree to maintain this stable dose for the duration of the study.

16. Medical use of cannabinoids and marijuana is permitted if the participant has a prescription, or (in states where over the counter cannabinoids including marijuana are legal) has a physician recommendation that cannabinoids are medically indicated over the counter that is clearly documented in the source file. Use must be stable for at least 4 weeks prior to baseline and for the duration of the study. They may not be used within 12 hours prior to cognitive or functional assessments.

Other Inclusion Criteria 17. Have one identified caregiver who has sufficient contact (approximately 10 hours a week or more) with direct contact, and has the ability to provide accurate information regarding the participant's cognitive and functional abilities and is willing to:

1. Attend all visits and report on participant's status
2. Oversee participant compliance with medication and study procedures
3. Provide informed consent and participate in the study assessments Note: In institutionalized settings (e.g., nursing homes or memory care facilities), a caregiver may be a staff member of the institutionalized setting or another individual (e.g., family member, family friend, hired professional caregiver) who fulfils the above criteria.

   -

   Exclusion Criteria:

   1. Risk of suicidal behaviour during the study as determined by the investigator's clinical assessment and/or C-SSRS (baseline version) as confirmed by the following:

a. Answers "Yes" on items 4, or 5 (C-SSRS-ideation) with the most recent episode occurring within the 2 months before screening or, b. Answers "Yes" to any of the 5 items (C-SSRS-behavior) with an episode occurring within the 12 months before screening 2. Any current primary psychiatric diagnosis (e.g., major depression, schizoaffective disorder, bipolar disorder) or severe psychiatric symptoms (e.g., hallucination, agitation or delusions) if, in the judgment of the investigator, the psychiatric disorder or symptom is likely to confound interpretation of treatment effect, affect cognitive assessment, or may impact the participants ability to complete the study.

3. Participants with history of schizophrenia or other chronic psychosis. 4. Any prior or on-going uncontrolled/unstable psychiatric disorder that could interfere with study assessments.

Medical Conditions 5. History or presence of clinically significant cardiovascular (e.g., untreated or unstable hypertension, clinically significant tachycardia), pulmonary, renal, hematologic, gastrointestinal (e.g., obstructive disorders [including conditions that may decrease GI motility, such as ulcerative colitis, intestinal atony, and myasthenia gravis]), endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the investigator, would jeopardize the safety of the participant or the validity of the study results.

6. History of ischemic stroke within 12 months prior to the screening visit, or any evidence of hemorrhagic stroke.

7. History of cerebral amyloid angiopathy, epilepsy, CNS neoplasm, or unstable thyroid function.

8. History or high risk of urinary retention (for male participants, includes PVR urine volume > 150 mL at screening; re-test is permitted when PVR urine volume is 151 through 175 mL at screening), gastric retention, or narrow-angle glaucoma.

9. Active biliary disease (e.g., symptomatic gallstones, cholangitis, biliary sphincter contraction, cholecystitis). A history of other biliary disease may be eligible and should be discussed with the medical monitor.

10. Participants with any of the following:

a. history of bladder stones b. history of recurrent urinary tract infections c. For male participants, serum prostate-specific antigen >10 ng/mL at screening d. For male participants, an IPSS score of 5 (i.e., "almost always") on items 1, 3, 5, or 6 e. For male participants, an IPSS score ≥ 9 for the sum of items 1, 3, 5, and 6 11. All grades of hepatic impairment (mild [Child-Pugh Class A], moderate [Child-Pugh Class B], and severe [Child-Pugh Class C]).

12. Participants with HIV with detectible viral load, HCV, cirrhosis, biliary duct abnormalities, hepatobiliary carcinoma, and/or active hepatic viral infections based on either medical history or LFT results.

13. History of irritable bowel syndrome (with or without constipation) or any serious constipation requiring treatment within the last 6 months.

14. History of allergy/hypersensitivity to any component (including excipients) of the study intervention or related compounds.

15. History of any of the following:

1. New York Heart Association Class II or greater congestive heart failure
2. Grade 2 or greater angina pectoris
3. Sustained ventricular tachycardia
4. Ventricular fibrillation
5. Torsades de pointes
6. Implantable cardiac defibrillator
7. Myocardial infarction within the 6 months prior to the screening visit.
8. Personal or family history of symptoms of long QT syndrome as evaluated by the investigator.

   16. Known acute infection or symptomatic illness within 2 weeks before screening; antigen or polymerase chain reaction local testing can be done at the discretion of the investigator. Rescreening can be permitted after the infection/illness is resolved and consultation with the medical monitor.

   17. Participation in another clinical study in which the participant received an experimental or investigational drug within 4 weeks before screening or has participated in more than 2 clinical studies in the 12 months prior to screening.

   18. Clinically significant abnormal finding on the physical or neurological examination, ECG, or clinical laboratory results at screening.

   19. Any significant pathological findings on historical brain MRI (prior to 14th infusion of Leqembi®) submitted at screening that could impact a participant's safety or interfere with study procedure, including, but not limited to: encephalomalacia, aneurysms, vascular malformations, infective lesions, evidence of any intracranial hemorrhage greater than 10 mm, more than 4 cerebral microbleeds, vasogenic edema, cerebral contusion or infection, more than 1 area of superficial siderosis, evidence of multiple lacunar infarcts (with an axial diameter of < 1.5 cm on neuroimaging) or stroke involving a major vascular territory, severe small vessel disease, or severe white matter disease as defined by a score of 3 on the Fazekas scale; space-occupying lesions or brain tumors (with the exception for meningiomas and arachnoid cysts < 1 cm in greatest diameter, which are permitted).

   20. Participants with any of the following:

a. history of unexplained syncope b. history of symptomatic orthostatic hypotension c. history of dysautonomia d. symptomatic orthostatic hypotension (symptomatic reduction of 20 mmHg or more in systolic blood pressure, and/or a symptomatic reduction of 10 mmHg or more in diastolic pressure) at screening. Asymptomatic orthostatic hypotension with a reduction of 20-30 mmHg in systolic blood pressure, and/or a reduction of 10 15 mmHg in diastolic pressure at screening may be eligible and should be discussed with the medical monitor.

21. History of medically significant bradycardia or heart rate < 50 bpm at screening.

Reproductive Status 22. Individuals who are pregnant, breastfeeding, or less than 3 months postpartum.

23. Any investigational therapy within 4 weeks prior to screening. 24. Prior exposure to X/T. 25. Currently taking or exposure to within 6 months prior to screening, a disease modifying anti- amyloid treatment for AD except Leqembi®.

26. Unable to taper and discontinue a concomitant medication that would preclude participation in this study (e.g., cannot stop potent anticholinergic or antihistamine medication).

27. No benzodiazepines may be taken within 12 hours prior to cognitive assessments (ADAS- Cog14, MMSE etc) unless taken regularly. If taken regularly, benzodiazepines must be taken at the same time interval prior to all cognitive assessments.

28. Recent history as defined as the past 3 months of receiving monoamine oxidase inhibitors, anticonvulsants (e.g., lamotrigine, divalproex), mood stabilizers (e.g., lithium), tricyclic antidepressants (e.g., imipramine, desipramine), or any other psychoactive medications except for as needed anxiolytics (e.g., lorazepam).

* Selective serotonin reuptake inhibitors and serotonin norepinephrine reuptake inhibitors taken at a stable dose for at least 12 weeks prior to screening may be permitted.
* MRTS (Mrazapine) or trazodone may be used as a hypnotic if started at least 8 weeks prior to screening.

  29. Inability to comply with restrictions and prohibited treatments as listed in Appendix 4.

Physical and Laboratory Test Findings 30. An eGFR of < 50 mL/min. 31. PSA ˃ 10 ng/ML at screening. 32. Elevations in hepatic transaminases at screening ≥ 3 × ULN for ALT and AST and/or bilirubin > 2 × ULN, unless in the context of Gilbert's syndrome.

33. Unstable hypertension or tachycardia as evidenced by:

1. Blood pressure of ≥ 150/100 mmHg (average of triplicate seated measures) at screening.
2. Heart rate of ≥ 100 bpm (average of triplicate seated measures) at screening. 34. Urine toxicology screen positive for phencyclidine, amphetamines, opiates, cocaine, or alcohol (clinically significant alcohol use in the opinion of the Investigator).

   35. Clinically significant abnormal finding on the physical examination, medical history, ECG (QTcF of > 450 msec in males and > 470 msec in females (as assigned at birth) ), or clinical laboratory results at screening.

   36. Vitamin B12 levels below LLN. Other Exclusion Criteria 37. Prisoners or participants who are involuntarily incarcerated. (Note: Under certain specific circumstances and only in countries where local regulations permit, a person who has been imprisoned may be included or permitted to continue as a participant. Strict conditions apply, and Sponsor approval is required).

   38. Participants with contraindications to the performance of brain MRI including cardiac pacemaker/defibrillator, ferromagnetic metal implants (e.g., in the skull and cardiac devices other than those approved as safe for use in MRI scanners).

   39. History of moderate-to-severe alcohol or substance use disorder within the past 2 years.

   40. If, in the opinion of the investigator and/or Sponsor/Medical Monitor, participant is unsuitable for enrollment in the study or participant has any finding that, in the view of the investigator and/or Sponsor/Medical Monitor, may compromise the safety of the participant or affect his/her ability to adhere to the protocol visit schedule or fulfil visit requirements.

   41. ApoE e4 homozygotes are not eligible. Subjects on anticoagulant therapy must have a stable dose for 4 weeks prior to screening and no history of ischemic or hemorrhagic stroke in the past 12 months or other neurological disorders.

   -

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Assess the safety and tolerability of X/T+X-EC compared with placebo in participants with Alzheimer's Disease currently treated with Lecanemab | Baseline to week 28 as there is a 4 week follow up period after End of Treatment
  Incidence of AEs/SAEs/AESIs/AEs leading to study intervention discontinuation, AEs leading to death through week 24.

SECONDARY OUTCOMES:
Quality of Life in Alzheimers Disease | Three different time points from Baseline to Week 24 will be assessed.
  Quality of Life-Alzheimer's Disease questionnaire is a measure to ensure the patient and caregiver construct validity and the measure focuses on aspects of life that are relevant to Alzheimer's Diseases. The total scoring sum is 13. The higher the score the better the participants Quality of Life. Questions will be answered as: poor, fair, good and excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Costell, MD, Principal Investigator — Neurology Office of South Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 20. Cobenfy (trospium-xanomeline). Package insert. Bristol-Myers Squibb Company; 2024.
- See also: Bristol- Myers Squibb — https://www.bms.com/